CLINICAL TRIAL: NCT00541450
Title: A Phase III Randomized, Active-Comparator (Pioglitazone) Controlled Clinical Trial to Study the Efficacy and Safety of Sitagliptin and MK0431A (A Fixed-Dose Combination Tablet of Sitagliptin and Metformin) in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Efficacy and Safety of Sitagliptin and MK0431A in Comparison to a Commonly Used Medication in Patients With Type 2 Diabetes (0431-068)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-068; 2007_501
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Sita/Met FDC (Experimental): In Phase A (Treatment Day 1 to Week 12), participants were administered 100 mg once daily (q.d.) of sitagliptin and matching placebo to 15 mg pioglitazone q.d. for 6 weeks followed by matching placebo to 30 mg pioglitazone for the next 6 weeks.
  In Phase B (Treatment Week 12-Week 40), participants were switched to the Sita/Met Fixed-Dose Combination (FDC) at a dose of 50/500 mg twice a day (b.i.d.), which was increased to 50/1000 mg b.i.d. over a period of 4 weeks; as well as matching placebo to 45 mg pioglitazone.
  Interventions: Drug: Comparator: sitagliptin phosphate (sitagliptin); Drug: sitagliptin phosphate (+) metformin hydrochloride; Drug: Matching placebo to pioglitazone
- Pioglitazone (Active Comparator): In Phase A (Treatment Day 1 up to Week 12), randomized participants in the pioglitazone group were administered 15 mg q.d. of pioglitazone and matching placebo to sitagliptin. At Week 6, participants were up-titrated to 30 mg pioglitazone q.d.
  In Phase B (Treatment Week 12 to Week 40), participants were administered 45 mg pioglitazone q.d.; as well as matching placebo to Sita/Met FDC (50/500 increased to 50/1000 b.i.d. after 4 weeks).
  Interventions: Drug: Comparator: pioglitazone; Drug: Matching placebo to sitagliptin; Drug: Matching Placebo to Sita/Met FDC

INTERVENTIONS:
Drug: Comparator: sitagliptin phosphate (sitagliptin) — sitagliptin 100 mg tablet q.d. orally for a 12-wk treatment period
  Other Names: MK0431, Januvia™
  Arms: Sita/Met FDC
Drug: sitagliptin phosphate (+) metformin hydrochloride — sitagliptin/metformin HCl (Sita/Met) 50/500 mg b.i.d. orally and then 50/1000 mg b.i.d. orally for a 28-wk treatment period
  Other Names: MK-0431A, Janumet™
  Arms: Sita/Met FDC
Drug: Comparator: pioglitazone — pioglitazone 15 mg tablet q.d. orally for 6 weeks, followed by 30 mg q.d orally for 6 weeks, followed by 45 mg q.d. orally, up to 40 weeks.
  Other Names: Actos®
  Arms: Pioglitazone
Drug: Matching placebo to pioglitazone — matching placebo to pioglitazone tablet q.d. orally, for a 40-wk treatment period.
  Participants were administered matching placebo the 15 mg pioglitazone q.d. orally for 6 weeks, followed by matching placebo to 30 mg pioglitazone q.d orally for 6 weeks, followed by matching placebo to 45 mg pioglitazone q.d. orally, up to 40 weeks.
  Arms: Sita/Met FDC
Drug: Matching placebo to sitagliptin — matching placebo to sitagliptin q.d., orally for a 12-wk treatment period.
  Arms: Pioglitazone
Drug: Matching Placebo to Sita/Met FDC — matching placebo to Sita/Met FDC - 50/500 mg b.i.d. for 4 weeks and then 50/1000 mg b.i.d. orally for a 28-wk treatment period (Week 12 to Week 40).
  Arms: Pioglitazone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sitagliptin and MK0431A in comparison to a commonly used medication in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 78 with type 2 diabetes mellitus
* Patient has not been on any antihyperglycemic agent (Insulin or oral) in the last 3 months

Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or a history of ketoacidosis
* Patient has previously been treated with sitagliptin or has previously been in a study using a DPP-4 inhibitor

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2008-01-15 (Actual); Primary Completion 2010-01-08 (Actual); Study Completion 2010-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Perez-Monteverde A, Seck T, Xu L, Lee MA, Sisk CM, Williams-Herman DE, Engel SS, Kaufman KD, Goldstein BJ. Efficacy and safety of sitagliptin and the fixed-dose combination of sitagliptin and metformin vs. pioglitazone in drug-naive patients with type 2 diabetes. Int J Clin Pract. 2011 Sep;65(9):930-8. doi: 10.1111/j.1742-1241.2011.02749.x. PMID 21849007

RESULTS

PARTICIPANT FLOW:
Groups:
- Sita/Met FDC: In Phase A (Treatment Day 1 up to Week 12), participants were administered 100 mg once daily (q.d.) of sitagliptin and matching placebo to pioglitazone.
  In Phase B (Treatment Week 12 to Week 40), participants that continued were switched to the Sita/Met Fixed-Dose Combination (FDC) at a dose of 50/500 mg twice a day (b.i.d.), which was increased to 50/1000 mg b.i.d. over a period of 4 weeks.
- Pioglitazone: In Phase A (Treatment Day 1 up to Week 12), participants in the pioglitazone group were administered 15 mg once daily (q.d.) of pioglitazone and matching placebo to sitagliptin. At Week 6, all participants were administered 30 mg q.d. pioglitazone.
  In Phase B (Treatment Week 12 to Week 40), participants that continued were administered 45 mg pioglitazone once daily (q.d.).
Period: Phase A
Arm/Group | Sita/Met FDC | Pioglitazone
Started | 244 | 248
Completed | 224 | 231
Not Completed | 20 | 17
Not completed — Adverse Event | 3 | 0
Not completed — Creatinine/CrCl -Increase in creatinine | 0 | 2
Not completed — Hyperglycemia | 0 | 1
Not completed — Lost to Follow-up | 6 | 4
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 7 | 7
Period: Phase B
Arm/Group | Sita/Met FDC | Pioglitazone
Started | 224 | 231
Completed | 187 | 200
Not Completed | 37 | 31
Not completed — Adverse Event | 6 | 6
Not completed — Hyperglycemia | 10 | 9
Not completed — Lost to Follow-up | 6 | 4
Not completed — Physician Decision | 4 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 3 | 3
Not completed — Withdrawal by Subject | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sita/Met FDC | Pioglitazone | Total
Number analyzed (Participants) | 244 | 248 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.5 (10.9) | 51.7 (10.1) | 51.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 100 | 192
  Male | 152 | 148 | 300

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (A1C) in the Sita/Met Fixed-Dose Combination (FDC) or Pioglitazone Groups at 40 Weeks
Description: The change in A1C, compared to baseline for the Sita/Met FDC and the pioglitazone groups at Week 40. A1C represents percentage of glycosylated hemoglobin.
Time Frame: Baseline to 40 weeks
Population: All randomized participants who (1) took at least one dose of study medication; i.e., sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12, and Sita/Met FDC or pioglitazone 45 mg q.d. for the Weeks 0-40 (Phase A and Phase B); and
  (2) had a baseline measurement and at least one on-treatment measurement for A1C.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Arm/Group | Sita/Met FDC | Pioglitazone
Number analyzed (Participants) | 218 | 222
percentage of glycosylated hemoglobin | -1.75 [-1.92 to -1.59] | -1.38 [-1.55 to -1.21]
Statistical Analysis 1: Comparison: Sita/Met FDC vs Pioglitazone; Test type: Superiority or Other; p = 0.002, ANCOVA; For Least Squares Mean, the ANCOVA model included a term for treatment and the baseline value as a covariate

2. Secondary Outcome: Change in 2-hour Postprandial Glucose (PMG) in the Sita/Met FDC or Pioglitazone Groups at 40 Weeks
Description: The change in PMG compared to baseline was measured using the Meal Tolerance Test (MTT) for the Sita/Met FDC and the pioglitazone groups at Week 40.
Time Frame: Baseline and 40 weeks
Population: All randomized participants who (1) took at least one dose of study medication; i.e., sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12, and Sita/Met FDC or pioglitazone 45 mg q.d. for the Weeks 0-40 (Phase A and Phase B); and
  (2) had a baseline measurement and at least one on-treatment measurement for PMG.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sita/Met FDC | Pioglitazone
Number analyzed (Participants) | 165 | 172
mg/dL | -90.3 [-99.6 to -81.0] | -69.1 [-78.2 to -60.0]
Statistical Analysis 1: Comparison: Sita/Met FDC vs Pioglitazone; Test type: Superiority or Other; p = 0.001, ANCOVA; For Least Squares Mean, the ANCOVA model included a term for treatment and the baseline value as a covariate

3. Primary Outcome: Change in Hemoglobin A1c (A1C) in Participants Treated With Sitagliptin or Pioglitazone at 12 Weeks
Description: The change in A1C compared to baseline was measured for the participants treated with sitagliptin or pioglitazone at Week 12. Sitagliptin was the only intervention administered to the Sita/Met FDC group during this phase. A1c represents percentage of glycosylated hemoglobin.
Time Frame: Baseline to 12 weeks
Population: All randomized participants who (1) took at least one dose of study medication; i.e., sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12; and (2) had a baseline measurement and at least one on-treatment measurement for A1C.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycosylated hemoglobin
Groups:
- Sitagliptin (Phase A): In Phase A (Treatment Day 1 up to Week 12), participants were administered 100 mg q.d. of sitagliptin or matching placebo.
- Pioglitazone (Phase A): In Phase A (Treatment Day 1 up to Week 12), participants in the Pioglitazone group were administered 15 mg q.d. of pioglitazone or matching placebo. At Week 6, participants were administered 30 mg q.d. pioglitazone.
Arm/Group | Sitagliptin (Phase A) | Pioglitazone (Phase A)
Number analyzed (Participants) | 231 | 240
percentage of glycosylated hemoglobin | -1.03 [-1.18 to -0.88] | -0.87 [-1.02 to -0.72]
Statistical Analysis 1: Comparison: Sitagliptin (Phase A) vs Pioglitazone (Phase A); Test type: Superiority or Other; ANCOVA; For Least Squares Mean, the ANCOVA model included a term for treatment and the baseline value as a covariate; Difference in LS Means = -0.16, 95% CI [-0.37 to 0.05]

4. Secondary Outcome: Change in 2-hour Postprandial Glucose (PMG) in Participants Treated With Sitagliptin or Pioglitazone at 12 Weeks
Description: The change in PMG compared to baseline was measured using the Meal Tolerance Test (MTT) for the participants treated with Sitagliptin or Pioglitazone at Week 12. Sitagliptin was the only intervention administered to the Sita/Met FDC group during this phase. To calculate Least Squares, the ANCOVA model included a term for treatment and the baseline value as a covariate.
Time Frame: Baseline to 12 weeks
Population: All randomized participants who (1) took at least one dose of study medication; i.e., sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12; and (2) had a baseline measurement and at least one on-treatment measurement for PMG.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin (Phase A) | Pioglitazone (Phase A)
Number analyzed (Participants) | 202 | 210
mg/dL | -52.8 [-62.4 to -43.3] | -50.1 [-59.4 to -40.7]

5. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) in the Sita/Met FDC or Pioglitazone Groups at 40 Weeks
Description: The change in FPG compared to baseline was measured for the Sita/Met FDC and the pioglitazone groups at Week 40.
Time Frame: Baseline and 40 weeks
Population: All randomized participants who (1) took at least one dose of study medication; i.e., sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12, and Sita/Met FDC or pioglitazone 45 mg q.d. for the Weeks 0-40 (Phase A and Phase B); and (2) had a baseline measurement and at least one on-treatment measurement for FPG.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sita/Met FDC | Pioglitazone
Number analyzed (Participants) | 219 | 226
mg/dL | -45.8 [-51.1 to -40.5] | -37.6 [-42.8 to -32.4]
Statistical Analysis 1: Comparison: Sita/Met FDC vs Pioglitazone; Test type: Superiority or Other; p = 0.030, ANCOVA; For Least Squares Mean, the ANCOVA model included a term for treatment and the baseline value as a covariate

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) in Participants Treated With Sitagliptin or Pioglitazone at 12 Weeks
Description: The change in FPG compared to baseline was measured for the participants treated with sitagliptin or pioglitazone at Week 12. Sitagliptin was the only intervention administered to the Sita/Met FDC group during this phase. To calculate Least Squares, the ANCOVA model included a term for treatment and the baseline value as a covariate.
Time Frame: Baseline to 12 weeks
Population: All randomized participants who (1) took at least one dose of study medication; i.e., sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12; and (2) had a baseline measurement and at least one on-treatment measurement for FPG.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin (Phase A) | Pioglitazone (Phase A)
Number analyzed (Participants) | 235 | 245
mg/dL | -26.6 [-31.7 to -21.5] | -28.0 [-33.0 to -23.0]

ADVERSE EVENTS:
Description: Participants that received at least one dose of study medication, which was sitagliptin or pioglitazone 15/30 mg q.d. for the Weeks 0-12 and Sita/Met FDC or pioglitazone 45 mg q.d. for the Weeks 0-40 were analyzed. The analyses for Week 0-40 did not include participants who discontinued from the study during Weeks 0-12.
Groups:
- Sitagliptin (Weeks 0-12): In Phase A (Treatment Day 1 up to Week 12), participants were administered 100 mg q.d. of sitagliptin or matching placebo to pioglitazone.
- Pioglitazone (Weeks 0-12): In Phase A (Treatment Day 1 up to Week 12), randomized participants in the pioglitazone group were administered 15 mg q.d. of pioglitazone or matching placebo to sitagliptin. At Week 6, all participants were up-titrated to 30 mg q.d. pioglitazone.
- Sita/Met FDC (Weeks 0-40): In Phase A (Treatment Day 1 up to Week 12), participants were administered 100 mg q.d. of sitagliptin or matching placebo to pioglitazone.
  In Phase B (Treatment Week 12-Week 40), participants were switched to the Sita/Met Fixed-Dose Combination (FDC) at a dose of 50/500 mg b.i.d., which was increased to 50/1000 mg b.i.d. over a period of 4 weeks.
- Pioglitazone (Weeks 0-40): In Phase A (Treatment Day 1 up to Week 12), randomized participants in the pioglitazone group were administered 15 mg q.d. of pioglitazone or matching placebo to sitagliptin. At Week 6, participants were up-titrated to 30 mg q.d.
  In Phase B (Treatment Week 12 -Week 40), participants were administered 45 mg q.d.
Arm/Group | Sitagliptin (Weeks 0-12) | Pioglitazone (Weeks 0-12) | Sita/Met FDC (Weeks 0-40) | Pioglitazone (Weeks 0-40)
Serious Adverse Events (participants affected / at risk) | 3/244 | 1/248 | 8/222 | 3/230
Other Adverse Events (participants affected / at risk) | 7/244 | 15/248 | 20/222 | 33/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (Weeks 0-12) (N=244) | Pioglitazone (Weeks 0-12) (N=248) | Sita/Met FDC (Weeks 0-40) (N=222) | Pioglitazone (Weeks 0-40) (N=230)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Infection parasitic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (Weeks 0-12) (N=244) | Pioglitazone (Weeks 0-12) (N=248) | Sita/Met FDC (Weeks 0-40) (N=222) | Pioglitazone (Weeks 0-40) (N=230)
Oedema peripheral (General disorders) | 0 (0) | 7 (7) | 2 (2) | 13 (15)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6) | 12 (14) | 12 (17)
Headache (Nervous system disorders) | 4 (4) | 4 (4) | 9 (13) | 12 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that an investigator and/or his/her colleagues may publish the results for their study site independently subsequent to the multicenter publication, or 24 months after completion of the study, whichever comes first. The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review.